CLINICAL TRIAL: NCT04523805
Title: Adapted Judo for Children With Autistic Spectrum Disorders
Acronym: AUTJUDO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Ramon Llull (Other)
Collaborators: Myriam Guerra (Unknown); Cristina Curto Luque (Unknown)
Responsible Party: Principal Investigator, Jose Morales, Principal Investigator, University Ramon Llull
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 01-autjudo
Record Dates: First submitted 2020-08-11; First posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Exercise intervention; Adapted judo intervention; GARS-3; TGMD-3
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Baseline data are collected at T1-Baseline, at the start of the programme and eight weeks later, scores are recorded for T2-Control, which represents a control period. During the control period, part of which includes the winter break from classes, the students not participate in any extracurricular physical activities, as their organised physical exercise is limited to their regular physical education classes at school. Between this second measurement and T3-Judo. T4-Follow up The judo sessions are performing in a large and well-ventilated space suitable for athletic activities in general and for judo in particular, such that the safety of the participants was maintained. Each participant is outfitted with a judogi (a traditional uniform consisting of a cotton jacket and trousers and a belt). The choice was made to include the control period at the start of the process because we did not have a control group willing to submit to all the measurements over the course of the project.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AUTJUDO-O1 (Experimental): The judo sessions are performing in a large and well-ventilated space suitable for athletic activities in general and for judo in particular, such that the safety of the participants was maintained. Each participant is outfitted with a judogi (a traditional uniform consisting of a cotton jacket and trousers and a belt).
  The sessions are 75 minutes in duration and were held once a week. Two judo teachers, with degrees in pedagogy and sports sciences and 7th and 6th degree black belts, respectively, led each session, and at least four volunteer judo instructors are present to lend support. The sessions are divided into warm-up, main exercise and cool-down activities. The instructional methodology apply the principles of gradual progression and the main exercise content of the sessions includes: different types of movements and falling techniques, ground control techniques, judo techniques and games.
  Interventions: Behavioral: Adapted judo programme

INTERVENTIONS:
Behavioral: Adapted judo programme — The judo sessions were 75 minutes in duration and were held once a week. Two judo teachers led each session, and at least four volunteer judo instructors were present to lend support. The sessions were divided into warm-up, main exercise and cool-down activities. The main exercise content of the sessions included:
  * Different types of movements and falling techniques (from walking in all directions to turning around, from stable movements to unstable movements).
  * Judo techniques and games (building up body contact with games, teaching simplified movements, essential judo movements) (blinded for review).
  * Ground control techniques and throws (gradually adding techniques to already known movements, scaffolding basic repetitive movements to assist in understanding to those more relevant for judo ).
  * Repetition of different forms of foundational directional movements (pulling, pushing, holding, lifting).

SUMMARY:
The project is aligned with one of the overall: To promote social inclusion and equal opportunities, encouraging participation in sport and physical activity. With this goal in mind, the following specific objectives for this project were established:

1. To develop an adapted judo programme for children with ASD.
2. To demonstrate the impact of the participation in adapted judo on the quality of life of people with ASD.
3. To validate instruments for use among the population with ASD.
4. To establish a set of coherent pedagogical principles that can be applied throughout the EU to ensure the effectiveness of adapted judo programmes for children with ASD.
5. To establish a coherent set of pedagogical principles to promote good habits in the participation in judo by children with ASD.
6. To consolidate and disseminate a systematic approach to adapted judo participation and competition for people with ASD around the EU.

Our hypothesis is that the participants will show improved behaviour after the adapted judo intervention

DETAILED DESCRIPTION:
The children were recruited via a number of associations of families with children with ASD and special education schools. All participants had been diagnosed with ASD according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition, (DSM-V). Individuals who had been advised against physical activity for medical reasons were excluded, as were those who had previously taken judo classes. The participants were invited to take part in the study voluntarily, and along with their parents were informed verbally and in writing as to the characteristics of the programme. Parents or legal guardians signed informed consent forms, and the children signed a consent document that explained the objectives and planned activities of the programme. The study was approved by the Research Ethics Committee of (blinded for review). All protocols applied in this research (including the management of the personal data of the participants) complied with the requirements specified in the Declaration of Helsinki of 1975 and its subsequent revisions.

The adapted judo programme is aimed at children of between 8 and 15 years of age who have been diagnosed with ASD and who being introduced to judo. All the project partners will contact institutions and organisations involved in the education of people with ASD in their respective localities and countries. The partners will explain the project and enlist the help of these institutions to recruit participants. All the study participants will be asked to sign an informed consent document that will be drafted in keeping with all applicable research ethics protocols, including a guarantee of the confidentiality of personal data and an assurance that participants can choose to abandon the study at any time.

The judo programme will be carried out over the course of two academic years (2020-21, 2021-22). The first school year will allow for pilot testing of the methods and point toward any necessary adaptations in the assessment techniques used. The design of this first phase will take into account prior experiences, expert input and information gleaned from focus groups in order to arrive at an initial proposal, which will then be subject to modification in accordance with results. The conclusions drawn from this initial experience will form the scientific and pedagogical basis for the definitive version of the programme.

The judo sessions will be offered in a large and well-ventilated space suitable for athletic activity in general and for judo in particular, such that the safety of the participants can be guaranteed. The judo equipment required for this project will include a tatami mat with a minimum surface area of 90 m2, made using high-density cushions that help prevent injuries and ensure that a wide range of activities can be carried out safely. Each participant will be outfitted with a judogui (a traditional uniform consisting of a cotton jacket and trousers and a belt that indicates the participant's level of technical skill).

The sessions will be an hour in length and will be held twice a week. Two instructors will lead each session, and at least four volunteers will have to be present to lend support. The sessions will be divided into three parts in accordance with the physiological principles of exercise: warm-up, main exercise and cool-down. The main content of the sessions will include:

* Judo analytical techniques and judo games
* Different types of movements and falling techniques.
* Ground control techniques and throws. The instruction methodology will always apply the principle of gradual progression, featuring practice to consolidate the concepts learned in the initial lessons before moving on to more complex material. Each participant will be allowed to progress at his or her own pace. Learning will be largely based on imitation and guided modelling of techniques.

This adapted judo programme for children with ASD will have broader scientific and pedagogical applications. Each project partner will be responsible for some data collection tasks. All the partners will gather pedagogical data throughout the process using a common methodology. Meanwhile, the scientific data will be gathered under stricter conditions by only some of the project partners. These data will then be handled and analysed by the research teams of the participating universities.

The judo sessions will be accompanied by the constant management and refining of the assessment and monitoring instruments that will be needed to gather the data that will inform the final results. Some of these instruments will be used pending a process of adaptation and validation for use with individuals with ASD, while others have already been tested and validated for use with this population. The following instruments will be administered during the programme:

* Test of Gross Motor Development (TGMD-2). Evaluates two components: a) Locomotor: Measures gross motor skills that require movements made with a fluid coordination (running, galloping, jumping with one foot, stride, jump with two feet slide). b) Object control: This subtest measures the gross motor skills that require efficiency when throwing, hitting and receiving (hitting a static ball, static jump, reception, shooting, throwing over the head and throwing below the head).
* Gilliam Autism Rating Scale (GARS-3). It consists of three subscales: Stereotypical behaviours, communication and social interaction. The instrument consists of 56 clearly stated items describing the characteristic behaviours of persons with autism. The items are grouped into six subscales: Restrictive/Repetitive Behaviours, Social Interaction, Social Communication, Emotional Responses, Cognitive Style, and Maladaptive Speech.
* Physical Activity Enjoyment Scale (PACES). It is a short questionnaire that asks about the degree of satisfaction when it comes to practicing physical activity.
* Battery ALPHA-FITNESS. It consists of the following variables: weight, height, body composition (abdominal perimeter, triceps sheet, subscapular fold), hand strength, leg strength, agility and aerobic endurance.
* Forms to record the participants' technical progress in judo (created for this study)

The pedagogical data will be collected by all the adapted judo instructors. In the collection of the research data, standard (blinded study) research protocols will be followed, and researchers will not be provided with information about the participants or the process carried out.

The two kinds of data described above will be handled differently. First, the pedagogical information will be subjected to qualitative analysis. These data will include expert opinion, the participants' level of satisfaction with the process and their degree of technical progress in judo. These qualitative data will be used to inform the drafting of the manuals for instructors of adapted judo for children with ASD, texts that will be produced within the framework of this project. Second, the scientific data will be subjected to quantitative analysis, including the use of more complex statistical methodology and of statistical analysis software. This quantitative analysis represents an opportunity validate some of the instruments applied in the study (PACES, ALPHA-FITNESS) for use among members of the autistic population. Also measured will be the performance of the participants in adapted judo competitions, the benefits of judo for individuals with ASD and the prevalence of injuries among participants in adapted judo.

Baseline data are collected at timepoint 1 (T1-Baseline), at the start of the programme and eight weeks later, scores are recorded for timepoint 2 (T2-Control), which represents a control period. During the control period, part of which includes the winter break from classes, the students not participate in any extracurricular physical activities, as their organised physical exercise is limited to their regular physical education classes at school. Between this second measurement and timepoint 3 (T3-Judo), The choice was made to include the control period at the start of the process because we did not have a control group willing to submit to all the measurements over the course of the project. In the absence of a control group, it was decided to take the second measurement after which the participants only took part in the compulsory physical education activities at their schools.

All descriptive data from the dependent variables are presented as mean ± standard deviation (SD). The normal distribution of each variable was checked with a Shapiro-Wilks test. In order to test the study hypotheses, comparisons between the four different timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ASD.

Exclusion Criteria:

* Clinical disability for physical activity

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Change from Pre-intervention in psycho-social and behavioural scores | Up to 16 weeks
  Gilliam Autism Rating Scale-Third Edition (GARS-3) scale (Gilliam, 2014). It includes 56 items describing characteristic behaviours of individuals with autism. The items are divided into six subscales: repetitive behaviours (RB), social interaction (SI), social communication (SC), emotional responses (ER), cognitive style (CS), and maladaptive speech (MS). Each item is scored on a four-point Likert-type scale (0=never observed; to 3=frequently observed), score indicates severity of autism-related behaviours and a lower value represents an improvement. The instrument can be administered by parents or caregivers in 5-10 minutes. It is based on the frequency of occurrence of each item under ordinary circumstances in a six-hour period. The raw score for each subscale was used. ), it should be noted that a low score indicates a decrease in the severity of the characteristics of children with ASD.
  Change= Pre-intervention (T2- control period) week 8- Post-intervention (T3-judo) week 16
Change from Pre-intervention in motor skills scores | Up to 16 weeks
  * Battery ALPHA-FITNESS. It obtains the following variables: weight, height, body composition (abdominal perimeter, triceps sheet, subscapular fold), hand strength, leg strength, agility and aerobic endurance. Scale will be reported (min 1-50) higher scores mean a better outcome.
  * Test of Gross Motor Development (TGMD-3). Evaluates two components: a) Locomotor: Measures gross motor skills that require movements made with a fluid coordination (running, galloping, jumping with one foot, stride, jump with two feet slide). b) Object control: This subtest measures the gross motor skills that require efficiency when throwing, hitting and receiving (hitting a static ball, static jump, reception, shooting, throwing over the head and throwing below the head). Scale will be reported (min 3-36) higher scores mean a better outcome.
  Change= Pre-intervention (T2- control period) week 8- Post-intervention (T3-judo) week 16

SECONDARY OUTCOMES:
Change from Baseline in psycho-social and behavioural scores | Up to 8 weeks
  Gilliam Autism Rating Scale-Third Edition (GARS-3) scale (Gilliam, 2014). It includes 56 items describing characteristic behaviours of individuals with autism. The items are divided into six subscales: repetitive behaviours (RB), social interaction (SI), social communication (SC), emotional responses (ER), cognitive style (CS), and maladaptive speech (MS). Each item is scored on a four-point Likert-type scale (0=never observed; to 3=frequently observed), score indicates severity of autism-related behaviours and a lower value represents an improvement. The instrument can be administered by parents or caregivers in 5-10 minutes. It is based on the frequency of occurrence of each item under ordinary circumstances in a six-hour period. The raw score for each subscale was used. ), it should be noted that a low score indicates a decrease in the severity of the characteristics of children with ASD.
  Change= Baseline (T1) week 0- Pre-intervention (T2) week 8
Change from Baseline in motor skills scores | Up to 8 weeks
  * Battery ALPHA-FITNESS. It obtains the following variables: weight, height, body composition (abdominal perimeter, triceps sheet, subscapular fold), hand strength, leg strength, agility and aerobic endurance. Scale will be reported (min 1-50) higher scores mean a better outcome.
  * Test of Gross Motor Development (TGMD-3). Evaluates two components: a) Locomotor: Measures gross motor skills that require movements made with a fluid coordination (running, galloping, jumping with one foot, stride, jump with two feet slide). b) Object control: This subtest measures the gross motor skills that require efficiency when throwing, hitting and receiving (hitting a static ball, static jump, reception, shooting, throwing over the head and throwing below the head). Scale will be reported (min 3-36) higher scores mean a better outcome.
  Change= Baseline (T1) week 0- Pre-intervention (T2) week 8

OTHER OUTCOMES:
Change from post-intervention in psycho-social and behavioural scores | Up to 24 weeks
  Gilliam Autism Rating Scale-Third Edition (GARS-3) scale (Gilliam, 2014). It includes 56 items describing characteristic behaviours of individuals with autism. The items are divided into six subscales: repetitive behaviours (RB), social interaction (SI), social communication (SC), emotional responses (ER), cognitive style (CS), and maladaptive speech (MS). Each item is scored on a four-point Likert-type scale (0=never observed; to 3=frequently observed), score indicates severity of autism-related behaviours and a lower value represents an improvement. The instrument can be administered by parents or caregivers in 5-10 minutes. It is based on the frequency of occurrence of each item under ordinary circumstances in a six-hour period. The raw score for each subscale was used. ), it should be noted that a low score indicates a decrease in the severity of the characteristics of children with ASD.
  Change=Post-intervention week 16- Follow up week 24
Change from post-intervention in motor skills scores | Up to 24 weeks
  * Battery ALPHA-FITNESS. It obtains the following variables: weight, height, body composition (abdominal perimeter, triceps sheet, subscapular fold), hand strength, leg strength, agility and aerobic endurance. Scale will be reported (min 1-50) higher scores mean a better outcome.
  * Test of Gross Motor Development (TGMD-3). Evaluates two components: a) Locomotor: Measures gross motor skills that require movements made with a fluid coordination (running, galloping, jumping with one foot, stride, jump with two feet slide). b) Object control: This subtest measures the gross motor skills that require efficiency when throwing, hitting and receiving (hitting a static ball, static jump, reception, shooting, throwing over the head and throwing below the head). Scale will be reported (min 3-36) higher scores mean a better outcome.
  Change=Post-intervention week 16- Follow up week 24
Level of Physical Activity Enjoyment | Up to 16 weeks
  -Physical Activity Enjoyment Scale (PACES). It is a short questionnaire that asks about the degree of satisfaction when it comes to practicing physical activity. Scale will be reported (min 0-20) higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Myriam Guerra-Balic, Dr, Study Chair — URamonLull
Locations (1):
- Jose Morales, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruiz JR, Castro-Pinero J, Espana-Romero V, Artero EG, Ortega FB, Cuenca MM, Jimenez-Pavon D, Chillon P, Girela-Rejon MJ, Mora J, Gutierrez A, Suni J, Sjostrom M, Castillo MJ. Field-based fitness assessment in young people: the ALPHA health-related fitness test battery for children and adolescents. Br J Sports Med. 2011 May;45(6):518-24. doi: 10.1136/bjsm.2010.075341. Epub 2010 Oct 19. PMID 20961915
- [Background] Karren, B. C. (2017). A Test Review: Gilliam, JE (2014). Gilliam Autism Rating Scale-Third Edition (GARS-3).
- [Background] Randall M, Egberts KJ, Samtani A, Scholten RJ, Hooft L, Livingstone N, Sterling-Levis K, Woolfenden S, Williams K. Diagnostic tests for autism spectrum disorder (ASD) in preschool children. Cochrane Database Syst Rev. 2018 Jul 24;7(7):CD009044. doi: 10.1002/14651858.CD009044.pub2. PMID 30075057
- [Background] Allen KA, Bredero B, Van Damme T, Ulrich DA, Simons J. Test of Gross Motor Development-3 (TGMD-3) with the Use of Visual Supports for Children with Autism Spectrum Disorder: Validity and Reliability. J Autism Dev Disord. 2017 Mar;47(3):813-833. doi: 10.1007/s10803-016-3005-0. PMID 28091840
- [Background] Latorre Roman PA, Garcia Pinillos F, Navarro Martinez AV, Izquierdo Rus T. Validity and reliability of Physical Activity Enjoyment Scale questionnaire (PACES) in children with asthma. J Asthma. 2014 Aug;51(6):633-8. doi: 10.3109/02770903.2014.898773. Epub 2014 Mar 24. PMID 24580370
- [Background] Teques P, Calmeiro L, Silva C, Borrego C. Validation and adaptation of the Physical Activity Enjoyment Scale (PACES) in fitness group exercisers. J Sport Health Sci. 2020 Jul;9(4):352-357. doi: 10.1016/j.jshs.2017.09.010. Epub 2017 Sep 29. PMID 32768128
- [Derived] Pierantozzi E, Morales J, Fukuda DH, Garcia V, Gomez AM, Guerra-Balic M, Carballeira E. Effects of a Long-Term Adapted Judo Program on the Health-Related Physical Fitness of Children with ASD. Int J Environ Res Public Health. 2022 Dec 13;19(24):16731. doi: 10.3390/ijerph192416731. PMID 36554612